CLINICAL TRIAL: NCT05077839
Title: Trifluridine/Tipiracil Combined With Oxaliplatin and Bevacizumab Versus XELOX Plus Bevacizumab in the First-line Treatment of Advanced Colorectal Cancer (TOBACO): a Randomized, Controlled, Phase II Study
Brief Title: Trifluridine/Tipiracil Combined With Oxaliplatin and Bevacizumab Versus XELOX Plus Bevacizumab in mCRC
Acronym: TOBACO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJMUCH-GI-CRC03
Record Dates: First submitted 2021-09-23; First posted 2021-10-14 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: First-line Treatment; Advanced Colorectal Cancer
Keywords: Trifluridine/tipiracil; first-line treatment; advanced colorectal cancer
MeSH Terms: interventions — trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): In the experimental group, the treatment regimen is trifluridine/tipiracil 35mg/m2 orally taken on d1-5 and d8-12, oxaliplatin 85mg/m2 and bevacizumab 5mg/kg intravenously infused on d1 and d15 every 4 weeks, up to 6 cycles. Then patients will be given trifluridine/tipiracil and bevacizumab maintenance treatment.
  Interventions: Drug: Trifluridine/Tipiracil
- control group (No Intervention): The control group was XELOX plus bevacizumab regimen, bevacizumab 7.5mg/kg, d1 oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, orally, bid (half an hour after breakfast and dinner), d1-14, every 3 weeks, up to 8 cycles. Then patients will be given capecitabine and bevacizumab maintenance treatment.

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Trifluridine/tipiracil was approved in the third-line treatment of advanced colorectal cancer. Its efficacy in the first-line treatment was unknown.
  Other Names: TAS-102
  Arms: experimental group

SUMMARY:
This is a two-group, parallel, randomized, standard-control phase II study comparing the safety and efficacy of trifluridine/tipiracil combined with oxaliplatin and bevacizumab versus XELOX plus bevacizumab in the first-line treatment of advanced colorectal cancer. This study was conducted in the Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Institute and Hospital.

Patients with advanced colorectal cancer will be randomly assigned (1:1) to trifluridine/tipiracil combined with oxaliplatin and bevacizumab (experimental group) or XELOX plus bevacizumab (control group) after signing informed consent. In this study, 184 patients will be enrolled, 92 patients will receive trifluridine/tipiracil combined with oxaliplatin and bevacizumab and 92 patients will receive standard therapy.

In the experimental group, the treatment regimen is trifluridine/tipiracil 35mg/m2 orally taken on d1-5 and d8-12, oxaliplatin 85mg/m2 and bevacizumab 5mg/kg intravenously infused on d1 and d15 every 4 weeks, up to 6 cycles. Then patients will be given trifluridine/tipiracil and bevacizumab maintenance treatment. Patients enrolled in this group could acquire trifluridine/tipiracil free of charge.

The control group was XELOX plus bevacizumab regimen, bevacizumab 7.5mg/kg, d1 oxaliplatin 130mg/m2, d1, capecitabine 1000mg/m2, orally, bid (half an hour after breakfast and dinner), d1-14, every 3 weeks, up to 8 cycles. Then patients will be given capecitabine and bevacizumab maintenance treatment.

Patients received regular and periodic reviews, with imaging evaluations every 8 weeks. Safety will be evaluated by AE and laboratory tests. All patients were followed up every 3 months until death according to the plan.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent.
2. Age ≥18.
3. Colonic adenocarcinoma confirmed histologically or histopathologically.
4. No previous chemotherapy for advanced colorectal cancer, or patients who had received adjuvant chemotherapy after radical resection and relapsed 12 months after the completion of adjuvant chemotherapy.
5. ECOG physical status score is 0 or 1.
6. There are measurable metastatic lesions according to RECIST version 1.1.
7. Appropriate organ function according to the following laboratory test values obtained within 7 days prior to use on Day 1 of Cycle 1:

   1. Hemoglobin value ≥9.0g/dL.
   2. Absolute neutrophil count ≥1,500/mm3 (≥1.5*109/L).
   3. Platelet count ≥100,000/mm3 (≥100*109/L).
   4. Total serum bilirubin ≤1.5* upper normal limit (ULN).
   5. Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤2.5* upper limit of normal value (ULN). If the abnormal liver function is due to liver metastasis, AST and ALT should be ≤5*ULN.
   6. Serum creatinine ≤1.5 times * upper limit of normal (ULN) or creatinine clearance ≥50ml/min.
8. The results of urine or serum pregnancy test within 7 days prior to treatment were negative. Women who are likely to become pregnant and men must agree to take adequate contraceptive measures during the study period until 6 months after the end of medication.
9. Survival is expected to be at least 3 months.
10. Willing and able to follow research procedures and visit plans.

Exclusion Criteria:

1. Has a serious illness or medical condition, including but not limited to the following:

   1. There are other active malignant tumors at the same time, excluding those that have not occurred for more than 5 years or carcinoma in situ that can be cured by adequate treatment.
   2. Known presence of brain metastases or leptomeningeal metastases.
   3. Systemic active infection (i.e., infection causes body temperature ≥38℃).
   4. Clinically significant intestinal obstruction, pulmonary fibrosis, renal failure, liver failure, or symptomatic cerebrovascular disease.
   5. Uncontrolled diabetes.
   6. Severe/unstable angina, New York Heart Association (NYHA) grade III or IV symptomatic congestive heart failure.
   7. Gastrointestinal bleeding of clinical significance.
   8. Known presence of human immunodeficiency virus (HIV) or acquired routine immunodeficiency syndrome (AIDS) -associated disease, or active hepatitis B or C.
   9. There are psychiatric disorders that may increase the risk associated with participating in the study or taking the study drugs, or may interfere with the interpretation of the study results.
2. Any of the following treatments were received within a specific time frame before the study drug was taken:

   1. Major surgery in the previous 4 weeks. (Major surgery refers to laparotomy, thoracotomy, and laparoscopic resection of internal organs. On-off of abdomen was excluded)
   2. Radiotherapy with extended field within the previous 4 weeks or radiotherapy with limited field within the previous 2 weeks.
   3. Any investigational drugs within the previous 4 weeks.
3. Presence of neurotoxicity of CTCAE grade 2 or above caused by adjuvant therapy.
4. Pregnant or lactating women.
5. The researcher did not consider it appropriate to enter the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
ORR | 48 months
  the rate of patients with PR and CR

SECONDARY OUTCOMES:
PFS | 48 months
  The time from the beginning of randomization to the time when the disease progresses or the patient dies from any cause.
OS | 48 months
  The time from the beginning of randomization to the time when the patient dies from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Ba, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No